CLINICAL TRIAL: NCT07301320
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Prospective, Investigator-Initiated Trial to Assess the Efficacy, Safety, and Pharmacokinetics of Epetraborole in Patients With Mycobacterium Abscessus Lung Disease: REBOUND Study
Brief Title: Epetraborole in Patients With Mycobacterium Abscessus Lung Disease
Acronym: REBOUND
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kevin Winthrop (Other)
Collaborators: AN2 Therapeutics, Inc (Industry)
Responsible Party: Sponsor-Investigator, Kevin Winthrop, Professor, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REBOUND Trial
Record Dates: First submitted 2025-12-22; First posted 2025-12-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Mycobacterium Abscessus Infection
Keywords: NTM; nontuberculous mycobacteria; Mycobacterium abscessus; M. abscessus; abscessus
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, the Sponsor, and the Funder will be blinded to treatment group assignments throughout the study. The Sponsor (e.g., clinical supply manager etc.) will have a designated randomization administrator who will maintain the randomization codes in accordance with standard operating procedures to ensure the blind is properly maintained. Only Sponsor personnel who require knowledge of treatment assignments will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- High Dose Epetraborole (Experimental): This arm is a daily treatment regimen of a 750mg oral dose of Epetraborole.
  Interventions: Drug: Epetraborole
- Low Dose Epetraborole (Experimental): This arm is a daily treatment regimen of a 500mg oral dose of Epetraborole.
  Interventions: Drug: Epetraborole
- High Dose Placebo (Placebo Comparator): This arm is a daily treatment regimen of a placebo, matching the high dose experimental arm.
  Interventions: Drug: Placebo
- Low Dose Placebo (Placebo Comparator): This arm is a daily treatment regimen of a placebo, matching the low dose experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epetraborole — High-dose intervention (750mg daily)
  Arms: High Dose Epetraborole
Drug: Epetraborole — Low-dose intervention (500mg daily)
  Arms: Low Dose Epetraborole
Drug: Placebo — Placebo intervention (matching the high-dose experimental intervention)
  Arms: High Dose Placebo
Drug: Placebo — Placebo intervention (matching the low-dose experimental intervention)
  Arms: Low Dose Placebo

SUMMARY:
This double-blind, randomized, placebo-controlled, parallel-group, multicenter, prospective, investigator-initiated trial will evaluate epetraborole (EBO) monotherapy in the treatment of adults with Mycobacterium abscessus complex (MABc) Lung Disease (LD) of mild to moderate severity. For this study, two EBO oral dose regimens will be studied in patients with MABc-LD, each compared to a placebo group (ie, 4 treatment groups): 500 mg daily and 750 mg daily. Detailed inclusion and exclusion criteria attempt to identify only those patients who have acceptable risks based upon the EBO preclinical findings, phase 1, phase 2, and Phase 3 experience; standard-of-care procedures; and the specified procedures of the study. Following receipt of informed consent, and a Screening period, eligible patients will be randomized to one of the 4 treatment groups to receive active or matched placebo EBO tablets for 84 days. Patients will be assessed for clinical and microbiological evidence of efficacy. At selected investigative sites, patients will undergo sparse PK sampling. Safety and tolerability will be determined by standard clinical and laboratory assessment, with oversight by a qualified and appropriately constituted Data Safety Monitoring Board (DSMB). Data collected during the study will be analyzed per a comprehensive Statistical Analysis Plan (SAP). The study will be registered on clinicaltrials.gov. The total duration of patient participation is approximately 6 months.

DETAILED DESCRIPTION:
Non-tuberculous mycobacterial lung disease (NTM-LD) is a chronic, debilitating disease that can cause significant morbidity and mortality, and reduces quality of life. The primary intervention to treat NTM-LD is antibiotic treatment to eliminate the causative pathogen and thereby prevent progression of NTM-associated lung destruction and respiratory compromise. Among NTM organisms causing pulmonary infection, Mycobacterium abscessus complex (MABc) LD requires particularly complicated, prolonged and onerous intravenous treatment regimens that are burdensome to patients. New therapeutic options, especially those that can be administered orally, represent a high unmet need.

Epetraborole (EBO), a boron-containing heterocycle also possessing amine and hydroxyl functional groups, blocks bacterial protein synthesis by inhibiting bacterial LeuRS. Epetraborole is active against Mycobacterium abscessus complex (MABc) organisms in vitro, including against isolates resistant to drugs commonly used to treat MABc-Lung Disease (LD) (e.g., clarithromycin and amikacin). To date, no clinical efficacy data are available for use of EBO in humans with MABc-LD. However, available nonclinical and PK data support the potential efficacy of EBO in MABc-LD. A Phase 1 human lung PK study in healthy volunteers showed that the exposure of EBO in alveolar (lung) macrophages, lung cells that are primarily infected with mycobacteria in NTM-LD, was approximately 5-fold higher than in plasma. EBO exposure in pulmonary epithelial lining fluid (ELF) is approximately 53% of that in plasma. Because NTM organisms may also be found in ELF, adequate EBO concentrations in that space are potentially important to achieve therapeutic success. Furthermore, PK/PD modeling data support the potential efficacy of EBO for treatment of MABc-LD. Since the EBO MIC90 for MABc isolates is ~256-fold lower than that observed for MAC isolates from the truncated EBO-301 Phase 2/3 study in treatment-refractory Mycobacterium avium complex lung disease, treatment outcomes in MABc-LD are expected to be favorable. The molecule therefore has the potential to address the unmet need in MABc-LD patients with limited treatment options.

For this study, two oral EBO dose regimens will be studied in patients with MABc-LD compared to placebo: 500 mg daily and 750 mg daily.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who are 18 years of age or older.
2. Willing and able to provide written informed consent.
3. Patients with MABc lung disease, meeting the following (a) Microbiological, (b) Clinical, (c) Radiographic

   a. Microbiological criteria: i. Documentation of at least 1 Pre-Study MABc-positive respiratory specimen (sputum or deep bronchial specimen) collected per standard of care within 6 months prior to signing the consent form.

   ii. At least 1 Screening MABc-positive expectorated or induced sputum sample. b. Clinical criteria: At least 2 of the following patient-reported clinical symptoms: i. Chest pain ii. Chronic cough iii. Coughing up blood iv. Fatigue v. Fever (documented by thermometer) vi. Mucus (sputum) production vii. Night sweats (drenching perspiration with no other obvious etiology, e.g. perimenopausal) viii. Poor appetite ix. Shortness of breath x. Weight loss (unintentional, more than 5% of usual weight in 6 to 12 months) c. Radiographic criteria: Non-contrast chest CT scan within 4 months prior to signing the ICF (Pre-Study chest CT) or within the Screening Period (Screening chest CT) with abnormalities consistent with MABc-LD based on local interpretation (e.g. Investigator or local radiologist).
4. Patients who, in the opinion of the investigator, will not require initiation of guideline-directed antibiotic therapy for treatment of MABc-LD within the next 6 months, and for whom a delay, in order for the subject to participate in a placebo-controlled clinical trial, is considered both reasonable and clinically acceptable.
5. Patients who are willing to comply with all the study activities and procedures throughout the duration of the study.

   1. Patients must agree to use an effective method of birth control, if applicable, as follows: Females of childbearing potential (FOCPs; defined in Appendix 1, Contraception Requirements) must commit to either sexual abstinence or use of at least 2 medically accepted, effective methods of birth control (defined in Contraception Requirements) from Screening through the EOS Visit
   2. Males who are sexually active with a FOCP must agree to use an effective barrier method of contraception (defined in Contraception Requirements) from Screening through the EOS Visit
6. Patients expected to survive with continued antimycobacterial therapy and appropriate supportive care from Screening through the LFU Visit, in the judgment of the Investigator.

Exclusion Criteria:

1. Patients with a presence of any suspected or confirmed disease or condition at Screening or the time of randomization that, in the opinion of the Investigator, may confound the assessment of symptom-based clinical response, including, but not limited to, the following:

   * Radiographic presence of cavitary disease (defined as a patient with one or more cavities >2 cm internal diameter)
   * Cystic fibrosis or other inherited disorders of airway ciliary dysfunction (e.g., primary ciliary dyskinesia)
   * Active allergic bronchopulmonary mycosis
   * Anticipated or planned lung surgery for treatment of MABc lung disease
   * Disseminated MABc infection, or other known or suspected non-pulmonary source of infection (e.g., infective endocarditis, osteomyelitis, meningitis, or urinary tract infection) requiring non-study antimicrobial therapy
   * Concomitant pulmonary infection requiring antimicrobial therapy, including infection caused by fungi, viruses, non-MABc mycobacteria (e.g., Mycobacterium tuberculosis, Mycobacterium avium intracellulare, Mycobacterium avium complex, Mycobacterium kansasii), or other bacteria (e.g., Pseudomonas aeruginosa, Staphylococcus aureus).

   Note: Patients with MABc lung disease and concomitant non-MABc lung infection requiring antimicrobial therapy must complete the antimicrobial treatment for the non-MABc infection prior to randomization. Patients with respiratory specimen cultures that contain growth of non-MABc organisms that are deemed by the Investigator to be respiratory tract colonizers and who do not require or receive specific antimicrobial therapy may remain eligible. The Investigator should discuss such cases with the Study Investigator prior to randomization and provide rationale for study eligibility in the source document.
2. Patients on brensocatib who have not been on a stable dose for at least 12 weeks.
3. Patients with active pulmonary malignancy (primary or metastatic) or any malignancy that required or would require chemotherapy or radiation therapy within 1 year prior to randomization through the LFU Visit.
4. Patients with creatinine clearance (CrCl) of <30 mL/min, as estimated by the Cockcroft-Gault formula, at Screening: Estimated CrCl (mL/min) = (140 - Age [years]) × Actual Body Weight [kg] × [0.85 if Female]) / (72 × Serum Creatinine [mg/dL]).
5. Patients with any of the following hematological findings:

   1. Hemoglobin <11.0 g/dL or <6.83 mmol/L.
   2. Donation of blood or plasma within 28 days prior to randomization; or symptomatic loss of blood or hemorrhage within 28 days prior to randomization.
   3. Pre-existing (inborn or acquired) disorder of hematopoiesis that could substantially worsen the effect of EBO on hemoglobin levels or potentially prevent hemoglobin recovery post cessation of treatment, for example, thalassemia, sickle cell disease, hemolytic anemia, Inherited bone marrow failure syndromes, myelodysplastic or myeloproliferative disorders, bone marrow transplantation
6. Patients with severe hemoptysis within 28 days prior to randomization, defined as >100 mL (approximately >7 tbsp blood) over any 24-hour period.
7. Patients with severe hepatic impairment, as evidenced by alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × upper limit of normal (ULN) or total bilirubin >2 × ULN, or clinical signs of cirrhosis or end-stage hepatic disease (e.g., ascites, hepatic encephalopathy).
8. Patients who are pregnant or breastfeeding.
9. Patients with a mean QT interval corrected using Fridericia's formula (QTcF) >500 msec based 12-lead ECG at Screening.
10. Patients with an immunodeficiency or an immunocompromised condition and risk for an opportunistic pulmonary infection, including:

    * History of lung transplantation
    * Known history of human immunodeficiency virus (HIV) infection plus either an active acquired immunodeficiency syndrome (AIDS)-defining illness in the past 12 months, or a known cluster of differentiation 4 (CD4) count <200/mm3 within the past 12 months
    * Neutropenia at Screening (absolute neutrophil count <1,000 neutrophils/mm3)
    * Use of immunosuppressive therapy at Screening that in the opinion of the Investigator may place the patient at risk for an opportunistic pulmonary infection, including transplant rejection medication and chronic systemic corticosteroids defined as ≥15 mg/day of prednisone or systemic equivalent for >4 weeks.
11. Patients with an anticipated start of new non-study antimycobacterial therapy to be administered at any time between Screening and EOT.
12. Patients who have participated in a clinical trial of an investigational agent within 30 days (or 5 half-lives, whichever is longer) prior to Screening.
13. Patients with any prior exposure to epetraborole.
14. Patients with any condition that, in the opinion of the Investigator, interferes with the ability to safely complete the study or adhere to study requirements, including the patient's inability or unwillingness to comply with all study assessments and visits.
15. Patients with hypersensitivity to any EBO excipient (e.g., microcrystalline cellulose, colloidal silicon dioxide, croscarmellose sodium, magnesium stearate, polyvinyl alcohol, titanium dioxide, polyethylene glycol, talc).
16. Patients with a history of eosinophilic interstitial pneumonitis

For eligibility purposes, vital signs, clinical laboratory tests, and ECGs may be repeated once if an abnormal result is observed at the initial reading during Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Response (NTM Symptom Evaluation Instrument) at Day 84 | Day 1 to Day 84
  Improvement in severity of at least 50% of the symptoms present at baseline and no deterioration in severity of symptoms present at baseline
Sputum culture conversion by Day 84 | Day 1 to Day 84
  Defined as 3 consecutive negative cultures one month apart without intervening or subsequent positives
Decrease in semi-quantitative sputum culture counts at Day 84 | Day 1 to Day 84
  Defined as improvement in sputum colony count category as defined by Griffith et al, 2015
Change from baseline in Quality of Life - Bronchiectasis (QOL-B) Respiratory Domain at Day 84 | Day 1 to Day 84
  QOL-B Domain scores range from 0 to 100, with higher scores indicating better health-related quality of life
Change from baseline in MACrO2 PRO at Day 84 | Day 1 to Day 84
  MACrO2 scores range from 0 to 100, with lower scores indicating better symptom-related quality of life
Sputum culture conversion by Day 56 | Day 1 to Day 56
  Defined as 2 consecutive negative cultures collected one month apart without intervening or subsequent positives

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGI-C) at Day 84 | Day 1 to Day 84
  The Patient Global Impression of Change Scale has a minimum value of 1 and a maximum value of 7. For this scale, higher scores indicate a worse outcome.
Patient Global Impression of Severity (PGI-S) at Day 84 | Day 1 to Day 84
  The Patient Global Impression of Severity Scale measures severity of a patient's overall status over the previous 7 days. The responses on this scale have a minimum value of 'None' and a maximum value of 'Very severe' related to severity. For this scale, higher scores ('Very severe') indicate a worse outcome.
Clinical Global Impression - Global Improvement Scale (CGI-I) at Day 84 | Day 1 to Day 84
  The Clinical Global Impression - Global Improvement Scale has a minimum value of 1 and a maximum value of 7, with 0 indicating the scale was not assessed. For this scale, higher scores indicate a worse outcome.
Clinical Global Impression - Severity (CGI-S) at Day 84 | Day 1 to Day 84
  The Clinical Global Impression - Severity of Illness Scale has a minimum value of 1 and a maximum value of 7, with 0 indicating the scale was not assessed. For this scale, higher scores indicate a worse outcome.
NTM Symptoms Scale (NTM-SS) Questionnaire at Day 84 | Day 1 to Day 84
  The Non-tuberculous Mycobacteria Symptoms Scale measures symptoms within the previous 7 days including respiratory, fatigue, temperature, appetite/weight, cognition/mood, and sleep. Questions on this scale have a minimum value of 'Never' and a maximum value of 'Always' related to the prevalence of symptoms. For this scale, higher scores ('Always') indicate a worse outcome.
Time to growth in liquid medium | Day 1 to Day 84
  Measured at Days 14, 28, 42, 56, and 84
Time to first negative sputum culture | Day 1 to Day 84
Proportion of patients with an on-treatment MABC isolate demonstrating decreasing sensitivity to EBO | Day 1 to Day 84
Sputum culture conversion by Day 84 | Day 1 to Day 84
  Defined as 2 consecutive negative cultures one month apart without intervening or subsequent positives

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Winthrop, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Cancer Institute. (2017). Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0. U.S. Department of Health and Human Services, National Institutes of Health, National Cancer Institute. https://doi.org/10.33329/ctcae.v5.0
- [Background] Bowman CJ, Becourt-Lhote N, Boulifard V, Cordts R, Corriol-Rohou S, Enright B, Erkman L, Harris J, Hartmann A, Hilpert J, Kervyn S, Mattson B, Morford L, Muller M, Powell M, Sobol Z, Srinivasan R, Stark C, Thompson KE, Turner KJ, Barrow P. Science-Based Approach to Harmonize Contraception Recommendations in Clinical Trials and Pharmaceutical Labels. Clin Pharmacol Ther. 2023 Feb;113(2):226-245. doi: 10.1002/cpt.2602. Epub 2022 May 5. PMID 35388453
- [Background] Kaneko T, Otoshi R, Sekine A, Baba T, Yamada C, Haga S, Tagami Y, Sawazumi T, Takemura T, Komatsu S, Hagiwara E, Ogura T. Drug-related pneumonitis caused by amikacin liposome inhalation suspension: One pathologically proven case and single-center experience. Respir Investig. 2024 Jul;62(4):513-516. doi: 10.1016/j.resinv.2024.04.003. Epub 2024 Apr 13. PMID 38615375
- [Background] Rimal B, Lippincott CK, Panthi CM, Xie Y, Keepers TR, Alley M, Lamichhane G. Efficacy of epetraborole against Mycobacteroides abscessus in a mouse model of lung infection. Antimicrob Agents Chemother. 2024 Aug 7;68(8):e0064824. doi: 10.1128/aac.00648-24. Epub 2024 Jul 17. PMID 39016592
- [Background] Li L, Henkle E, Youngquist BM, Seo S, Hamed K, Melnick D, Lyon CJ, Jiang L, Zelazny AM, Hu TY, Winthrop KL, Ning B. Serum Cell-Free DNA-based Detection of Mycobacterium avium Complex Infection. Am J Respir Crit Care Med. 2024 May 15;209(10):1246-1254. doi: 10.1164/rccm.202303-0401OC. PMID 38190702
- [Background] Griffith DE, Adjemian J, Brown-Elliott BA, Philley JV, Prevots DR, Gaston C, Olivier KN, Wallace RJ Jr. Semiquantitative Culture Analysis during Therapy for Mycobacterium avium Complex Lung Disease. Am J Respir Crit Care Med. 2015 Sep 15;192(6):754-60. doi: 10.1164/rccm.201503-0444OC. PMID 26068042
- [Background] Eckburg PB, Clarke D, Long J, et al. 2022. Tolerability and pharmacokinetics of oral epetraborole at the predicted therapeutic dosage for Mycobacterium avium complex (MAC) lung disease: a phase 1b dose-ranging and food effect study. In ID week. Washington DC
- [Background] Griffith DE, Daley CL. Treatment of Mycobacterium abscessus Pulmonary Disease. Chest. 2022 Jan;161(1):64-75. doi: 10.1016/j.chest.2021.07.035. Epub 2021 Jul 24. PMID 34314673
- [Background] Daley CL, Iaccarino JM, Lange C, Cambau E, Wallace RJ Jr, Andrejak C, Bottger EC, Brozek J, Griffith DE, Guglielmetti L, Huitt GA, Knight SL, Leitman P, Marras TK, Olivier KN, Santin M, Stout JE, Tortoli E, van Ingen J, Wagner D, Winthrop KL. Treatment of Nontuberculous Mycobacterial Pulmonary Disease: An Official ATS/ERS/ESCMID/IDSA Clinical Practice Guideline. Clin Infect Dis. 2020 Aug 14;71(4):e1-e36. doi: 10.1093/cid/ciaa241. PMID 32628747
- [Background] Strnad L, Winthrop KL. Treatment of Mycobacterium abscessus Complex. Semin Respir Crit Care Med. 2018 Jun;39(3):362-376. doi: 10.1055/s-0038-1651494. Epub 2018 Aug 2. PMID 30071551
- [Background] Diel R, Ringshausen F, Richter E, Welker L, Schmitz J, Nienhaus A. Microbiological and Clinical Outcomes of Treating Non-Mycobacterium Avium Complex Nontuberculous Mycobacterial Pulmonary Disease: A Systematic Review and Meta-Analysis. Chest. 2017 Jul;152(1):120-142. doi: 10.1016/j.chest.2017.04.166. Epub 2017 Apr 28. PMID 28461147